CLINICAL TRIAL: NCT03941353
Title: Care Pathways for Benchmarking on Fragile Hip Fractures Rapid Recovery
Status: Completed | Type: Observational
Sponsor: European Pathway Association (Other)
Collaborators: KU Leuven (Other)
Responsible Party: Principal Investigator, Dr. Kris Vanhaecht, Professor in Healthcare Quality Management, European Pathway Association
Other Study IDs: CP4FHF
Record Dates: First submitted 2019-05-06; First posted 2019-05-07 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Quality Improvement; Hip Fractures
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Usual care — Benchmark study with retrospective patient analysis evaluating the actual care patients with a fragile hip fracture receive

SUMMARY:
The aim of this project is to build an international community of centers of excellence in the care for Fragile Hip Fracture Rapid Recovery patients. These centers of excellence will benchmark and share their expertise and experiences based on clinical and managerial data. In project is designed in five different phase:

Phase 1: literature review: identifying relevant key interventions and indicators Phase 2: expert panel: expert panel for teams, management and policy makers Phase 3: data collection: collection managerial data through retrospective patient record analysis on clinical indicators Phase 4: statistical data analysis: data input, validation and statistical analysis Phase 5: feedback and knowledge sharing: feedback report with anonymous benchmarking and knowledge sharing of the results.

ELIGIBILITY:
Inclusion Criteria:

* Trauma related non-elective admission for hip fracture;
* Minimum age of 65 years;
* The following hip fractures are included: Femoral neck, femoral head, trochanteric and subtrochanteric fractures;
* Discharged or deceased before May 30th of 2019

Exclusion Criteria:

* Hip fracture is not the main reason for admission to emergency room;
* Additional ipsilateral fractures;
* Hip fracture resulting from in-hospital fall that occurred in the hospital where the patient receives hip fracture care.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patient admitted with a proximal femur fracture
Sampling Method: Non-Probability Sample
Enrollment: 298 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-06-27 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Performance on quality indicators at patient level (Quality of Care and patient satisfaction) for patients admitted with a fragile hip fracture. | through study completion, an average of 1 year
  This study evaluates quality indicators at patient level as defined by the expert panel to determine appropriateness of fragile hip fracture indicators. The indicators will cover the pre-operative, peri-operative and post-operative care process. The data will be selected out of the patient record. Based on the expert panel quality of care is measured by time to surgery, information on pre-fall cognitive status, information on pre-fall mobility status, fasting time, administration of carbohydrate loading, administration of cortical steriods, use of tranexamic acid, urinary catheterization, administration of pain medication, time to post operative surgeon note for care team, time of drain duration, type of anesthesia, measurement of haemoglobin, mobilisation post-operative, following of pain protocol, plan for discharge, nutrition supplementation. he study is limited to the period in which the patients are hospitalized. No data is gathered before or after hospitalization.

CONTACTS AND LOCATIONS:
Locations (1):
- KU Leuven, Leuven, Belgium